CLINICAL TRIAL: NCT00523237
Title: Raltegravir Substitution for Enfuvirtide in Patients Suffering From Injection Site Reactions (ISRs): The Raleve Pilot Study
Brief Title: RAL-eve Study: Raltegravir Substitution Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAL-eve study; NCT00627939 (obsolete NCT alias)
Record Dates: First submitted 2007-08-29; First posted 2007-08-31 (Estimated); Results first posted 2011-10-28 (Estimated); Last update posted 2011-11-02 (Estimated); Status verified 2011-10

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Raltegravir — 400 mg Twice daily for 24 weeks
  Other Names: Isentress

SUMMARY:
The purpose of this study is to:

* Provide raltegravir to subjects with HIV and an undetectable viral load who are experiencing injection site reactions (ISR) to Enfuvirtide,
* Monitor the safety and efficacy of raltegravir, and
* Assess the change in quality of life in patients who have switched from Enfuvirtide to raltegravir

DETAILED DESCRIPTION:
We enrolled virologically suppressed HIV-1 infected patients with injection site reactions for a switch from enfuvirtide to raltegravir. At baseline, enfuvirtide was switched to raltegravir without additional changes to the antiretroviral regimen allowed. Viral load, T-cells, and toxicity were evaluated at baseline, 2, 4, 12 and 24 weeks. Adherence and injection site reactions were evaluated at baseline, 4, 12 and 24 weeks. The single-copy assay was used to measure HIV RNA levels at screening, baseline and at 12 and 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 infection, as documented by any licensed ELISA test kit and confirmed by Western blot at any time prior to study entry.
2. ART for at least 6 months prior to study entry with a regimen that includes enfuvirtide.
3. Self-defined infusion site reaction to enfuvirtide (usually will be painful inflammatory nodules)
4. No change in ART regimen for at least 3 months prior to study entry.
5. CD4+ cell count >50/mm3 at screening (obtained within 60 days prior to study entry).
6. Documentation of HIV-1 RNA below the limit of quantification of an ultrasensitive assay
7. All HIV-1 RNA levels obtained within 6 months prior to study entry are below the limits of quantification on all tests, except as explained above in section 4.1.6 for a single detectable viral load of <50 copies but <200 copies in last 6 months.
8. Laboratory values obtained within 60 days prior to entry:

   * Absolute neutrophil count (ANC) >750/mm3
   * Hemoglobin >9.0 g/dL for female subjects and>10.0 g/dL for male subjects
   * Platelet count >50,000/mm3
   * Calculated creatinine clearance (CrCl) >30 mL/min, as estimated by the Cockcroft-Gault equation*
   * AST (SGOT), ALT (SGPT), and alkaline phosphatase <5 x ULN
   * Total bilirubin <2.5 x ULN. If the subject is taking an indinavir- or atazanavir-containing regimen at the time of screening, total bilirubin <5 x ULN is acceptable.
9. For females of reproductive potential will need a negative serum or urine pregnancy test within 48 hours prior to entry.
10. Men and women age >18 years.
11. Ability and willingness of subject to provide informed consent.

Exclusion Criteria:

1. Unstable clinical condition, such as unstable cardiac disease, or cancer requiring ongoing chemotherapy or radiation therapy, or other medical condition which, in the opinion of the investigator, would preclude a subject from safely undergoing study procedures.
2. Breast-feeding or pregnancy.
3. An opportunistic infection within 60 days prior to entry.
4. Known allergy/sensitivity or any hypersensitivity to components of study drug(s) or their formulation.
5. Active drug or alcohol use or dependence that, in the opinion of the Protocol Director, would interfere with adherence to study requirements.
6. Receipt of a non-HIV vaccination within 30 days prior to study entry or plan for receipt of vaccination during the study.
7. Plan to change the background ART within 24 weeks after study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-10; Primary Completion 2009-03 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew R Zolopa, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Result] Grant PM, Palmer S, Bendavid E, Talbot A, Slamowitz DC, Cain P, Kobayashi SS, Balamane M, Zolopa AR. Switch from enfuvirtide to raltegravir in virologically suppressed HIV-1 infected patients: effects on level of residual viremia and quality of life. J Clin Virol. 2009 Dec;46(4):305-8. doi: 10.1016/j.jcv.2009.09.025. Epub 2009 Oct 12. PMID 19819183

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fourteen patients, all men, were enrolled.
Pre-assignment Details: All screened patients were enrolled into the study
Groups:
- Raltegravir: 400 mg twice daily
Period: Overall Study
Arm/Group | Raltegravir
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Raltegravir
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 56 (56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 14
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Patients Who Maintain a Viral Load < 50 Copies/ml After Being Switched From Enfuvirtide to Raltegravir
Description: evaluate the percent of patients with viral load of <50 copies at week 24 of study after being switched from enfuvirtide to raltegravir
Time Frame: 24 weeks
Population: With expected man baseline residual viremia of 5 copies/ml and predicted standard deviation of 3 in change of residual viremia, our study was predicted to have 80% power to detect a difference of 2.5 copies/ml in residual viremia with =0.05.
Measure: Number; unit: percentage
Groups:
- Enfuvirtide Switch to Raltegravir Arm: patients were switched from Enfuvirtide to Raltegravir
Arm/Group | Enfuvirtide Switch to Raltegravir Arm
Number analyzed (Participants) | 14
percentage | 86

ADVERSE EVENTS:
Arm/Group | Raltegravir
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes